CLINICAL TRIAL: NCT04153656
Title: Impact of Spiritual Flow Compendium on Nurse Wellbeing
Brief Title: Spiritual Flow and Nurse Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Health Ohio (Other)
Collaborators: St. Elizabeth Youngstown Hospital (Unknown)
Responsible Party: Principal Investigator, C. Michael Dunham, Research Investigator, Mercy Health Ohio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-022
Record Dates: First submitted 2019-10-18; First posted 2019-11-06 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Burnout, Professional
Keywords: Burnout; Nurse wellbeing; Physician burnout; Nurse burnout
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurses (Other): Subjects will be asked to commit to reading and studying Spiritual Flow.
  Interventions: Other: Reading and studying Spiritual Flow

INTERVENTIONS:
Other: Reading and studying Spiritual Flow — The Wellbeing Inventory will be administered to subjects and they will be compensated upon completion of the survey. Two months after the first survey, the Wellbeing Inventory will be administered to subjects and they will be compensated upon completion of the survey.

SUMMARY:
The investigators hypothesize that wellbeing scores following the study of Spiritual Flow, when compared to taking the survey before receiving Spiritual Flow, will increase. Pre- and post-Spiritual Flow assessments will include wellbeing, nonstress, and positive affect scores. The investigators also hypothesize that several subjects will have found that Spiritual Flow increased their level of inspiration and peacefulness.

DETAILED DESCRIPTION:
Multiple investigations document substantial concerns relative to emotional exhaustion, burnout, and job dissatisfaction in nurse and physician cohorts. Physician research has demonstrated considerable pervasiveness of emotional exhaustion, emotional hardening, burnout, depression, suicidal ideation, and fatigue. Emotional exhaustion, a risk for burnout, has also been found to be substantial in nurses in the United States. Surveys have indicated that 20-35% of hospital-based nurses have expressed the intent to leave their current job in the near future.

There is no single study that includes United States physicians and nurses and then provides subset analyses that compare physician to nurse burnout in the same healthcare environment. However; comparisons, although with limited conclusions, can be based on separate studies. The 33% burnout proportion in a nurse study is lower than the 40-55% proportion described in physician investigations; however, substantial in both. Data from a systematic review of intensive care unit professionals indicates that the emotional exhaustion proportion for nurses has a mean of 32% (5 studies) and for physicians is 25% (1 study). Physician emotional exhaustion scores (22-25) are similar to the 2 studies describing nurse emotional exhaustion scores (24). The proportions of depression for physicians have been reported to be similar to those for nurses. The job dissatisfaction proportion for physicians has been shown to be comparable to those for nurses. The investigators found 3 recent Middle Eastern studies demonstrating that physician and nurse burnout proportions and high emotional exhaustion proportions were similar when the physicians and nurses worked in the same healthcare environment.

In the past, the authors designed an 11-item nurse and physician survey, the St. Elizabeth Youngstown Hospital Wellbeing Inventory. The 4 positive affect items (restful sleep, energetic, alert, and enthusiastic) were each ranked as 1) very slightly or none at all, 2) a little, 3) moderately, 4) quite a bit, or 5) extremely. The positive affect score was the sum of the ratings for these 4 items. The 7 negative affect items (irritation, nervousness, overreaction, tension, feeling overwhelmed, feeling that people were too demanding, and feeling drained) were each ranked, using reversed coding, as 5) very slightly or none at all, 4) a little, 3) moderately, 2) quite a bit, or 1) extremely. The positive affect score was the sum of the ratings for the 4 positive affect items (range 4-20). The nonstress score was the sum of the reverse-scored ratings for the 7 negative affect items (range 7-35). The wellbeing score was the sum of the positive affect and nonstress scores (range 11-55). The Wellbeing Inventory has been demonstrated to be valid, according to psychometric properties, and can be considered to be most relevant to United States nurses and physicians working in a hospital-trauma center environment.

The content of Spiritual Flow: Pathways to Proficient Patient Care and Nurse & Physician Wellbeing (available on Amazon.com) came directly from Authentic Sports: The 7 Pathways to Peak Performance, second edition, written by Bill Lefko and Daniel Baird. Authentic Sports is a guide for enhancing sports performance and increasing joy while playing sports. Guidance is provided using spiritual principles as they affect various sporting activities. Multiple sport vignettes are included throughout the guide to complement and illustrate the principles as they are being presented. The essence of each principle is virtually identical whether one is discussing sports activities; waitressing; machine shop working; or providing patient care. Accordingly, virtually all of the statements in Spiritual Flow are identical to that printed in Authentic Sports and written by Bill Lefko and Daniel Baird. C. Michael Dunham, MD changed a small percent of the language such that physicians and nurses reading the compendium would better relate to the content and better understand the principles that were presented in Authentic Sports. The sports vignettes were deleted to shorten the reading duration for time-limited physicians and nurses.

In chapter 9 of Spiritual Flow are guided meditations to assist nurses and physicians in enhancing mindfulness experiences during patient care activities. Mindfulness is an attitudinal expression of receptive awareness, wherein there is a distinction made between an experience occurring in the present moment and associated thoughts and interpretations about that experience. The thinking process itself is observed with all thoughts being treated as equal in value, without attraction or rejection. In two investigations that consisted of physicians and nurses, a high mindfulness score was associated with less stress, greater wellbeing, and a positive emotional tone among subjects. Mindfulness training has been associated with reductions in stress or burnout risk in literature reviews focusing on nurses or physicians and in studies that include nurses and physicians.

ELIGIBILITY:
Inclusion Criteria:

* Nurses (registered, practitioner, and anesthetist), employed at St. Elizabeth Youngstown Trauma Center, Mercy Health, will be welcomed to participate in the study.

Exclusion Criteria:

* Non-nurse employees of St. Elizabeth Youngstown Trauma Center, Mercy Health

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
St. Elizabeth Youngstown Hospital Wellbeing Inventory - Wellbeing score | Up to 6 months
  Change in wellbeing scores following the study of Spiritual Flow, when compared to taking the survey before receiving Spiritual Flow. The wellbeing score was the sum of the positive affect and nonstress scores (range 11-55).

SECONDARY OUTCOMES:
St. Elizabeth Youngstown Hospital Wellbeing Inventory - Nonstress score | Up to 6 months
  Nonstress score pre- and post-Spiritual Flow assessments. The nonstress score was the sum of the reverse-scored ratings for the 7 negative affect items (range 7-35).
St. Elizabeth Youngstown Hospital Wellbeing Inventory - Positive affect score | Up to 6 months
  Positive affect score pre- and post-Spiritual Flow assessments. The 4 positive affect items (restful sleep, energetic, alert, and enthusiastic) were each ranked as 1) very slightly or none at all, 2) a little, 3) moderately, 4) quite a bit, or 5) extremely. The positive affect score was the sum of the ratings for these 4 items (range 4-20).

CONTACTS AND LOCATIONS:
Overall Officials: C. Michael Dunham, MD, Principal Investigator — St. Elizabeth Youngstown Hospital
Locations (1):
- St. Elizabeth Youngstown Hospital, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon individual request; there are no individual subject traits on the surveys; only survey response results will be made available
Time Frame: Data will become available starting 6 months after publication
Access Criteria: Data will be provided upon request by emailing the principal investigator

REFERENCES:
- [Background] Dyrbye LN, Satele D, Sloan J, Shanafelt TD. Utility of a brief screening tool to identify physicians in distress. J Gen Intern Med. 2013 Mar;28(3):421-7. doi: 10.1007/s11606-012-2252-9. Epub 2012 Nov 6. PMID 23129161
- [Background] Dyrbye LN, West CP, Satele D, Boone S, Tan L, Sloan J, Shanafelt TD. Burnout among U.S. medical students, residents, and early career physicians relative to the general U.S. population. Acad Med. 2014 Mar;89(3):443-51. doi: 10.1097/ACM.0000000000000134. PMID 24448053
- [Background] Brazeau CM, Shanafelt T, Durning SJ, Massie FS, Eacker A, Moutier C, Satele DV, Sloan JA, Dyrbye LN. Distress among matriculating medical students relative to the general population. Acad Med. 2014 Nov;89(11):1520-5. doi: 10.1097/ACM.0000000000000482. PMID 25250752
- [Background] Poghosyan L, Clarke SP, Finlayson M, Aiken LH. Nurse burnout and quality of care: cross-national investigation in six countries. Res Nurs Health. 2010 Aug;33(4):288-98. doi: 10.1002/nur.20383. PMID 20645421
- [Background] Vahey DC, Aiken LH, Sloane DM, Clarke SP, Vargas D. Nurse burnout and patient satisfaction. Med Care. 2004 Feb;42(2 Suppl):II57-66. doi: 10.1097/01.mlr.0000109126.50398.5a. PMID 14734943
- [Background] Chang EM, Bidewell JW, Huntington AD, Daly J, Johnson A, Wilson H, Lambert VA, Lambert CE. A survey of role stress, coping and health in Australian and New Zealand hospital nurses. Int J Nurs Stud. 2007 Nov;44(8):1354-62. doi: 10.1016/j.ijnurstu.2006.06.003. Epub 2006 Aug 9. PMID 16901488
- [Background] Lindqvist R, Smeds Alenius L, Griffiths P, Runesdotter S, Tishelman C. Structural characteristics of hospitals and nurse-reported care quality, work environment, burnout and leaving intentions. J Nurs Manag. 2015 Mar;23(2):263-74. doi: 10.1111/jonm.12123. Epub 2013 Sep 19. PMID 24047463
- [Background] Poncet MC, Toullic P, Papazian L, Kentish-Barnes N, Timsit JF, Pochard F, Chevret S, Schlemmer B, Azoulay E. Burnout syndrome in critical care nursing staff. Am J Respir Crit Care Med. 2007 Apr 1;175(7):698-704. doi: 10.1164/rccm.200606-806OC. Epub 2006 Nov 16. PMID 17110646
- [Background] Embriaco N, Papazian L, Kentish-Barnes N, Pochard F, Azoulay E. Burnout syndrome among critical care healthcare workers. Curr Opin Crit Care. 2007 Oct;13(5):482-8. doi: 10.1097/MCC.0b013e3282efd28a. PMID 17762223
- [Background] Chuang CH, Tseng PC, Lin CY, Lin KH, Chen YY. Burnout in the intensive care unit professionals: A systematic review. Medicine (Baltimore). 2016 Dec;95(50):e5629. doi: 10.1097/MD.0000000000005629. PMID 27977605
- [Background] Mealer ML, Shelton A, Berg B, Rothbaum B, Moss M. Increased prevalence of post-traumatic stress disorder symptoms in critical care nurses. Am J Respir Crit Care Med. 2007 Apr 1;175(7):693-7. doi: 10.1164/rccm.200606-735OC. Epub 2006 Dec 21. PMID 17185650
- [Background] Abdo SA, El-Sallamy RM, El-Sherbiny AA, Kabbash IA. Burnout among physicians and nursing staff working in the emergency hospital of Tanta University, Egypt. East Mediterr Health J. 2016 Mar 15;21(12):906-15. doi: 10.26719/2015.21.12.906. PMID 26996364
- [Background] Alqahtani AM, Awadalla NJ, Alsaleem SA, Alsamghan AS, Alsaleem MA. Burnout Syndrome among Emergency Physicians and Nurses in Abha and Khamis Mushait Cities, Aseer Region, Southwestern Saudi Arabia. ScientificWorldJournal. 2019 Feb 18;2019:4515972. doi: 10.1155/2019/4515972. eCollection 2019. PMID 30906233
- [Background] Hamdan M, Hamra AA. Burnout among workers in emergency Departments in Palestinian hospitals: prevalence and associated factors. BMC Health Serv Res. 2017 Jun 15;17(1):407. doi: 10.1186/s12913-017-2356-3. PMID 28619081
- [Background] Dunham CM, Burger AL, Hileman BM, Chance EA. Psychometric properties of the St. Elizabeth Youngstown hospital wellbeing inventory and non-burnout inventory for physicians and nurses. BMC Psychol. 2019 Jun 17;7(1):36. doi: 10.1186/s40359-019-0316-x. PMID 31208464
- [Background] Perlman DM, Salomons TV, Davidson RJ, Lutz A. Differential effects on pain intensity and unpleasantness of two meditation practices. Emotion. 2010 Feb;10(1):65-71. doi: 10.1037/a0018440. PMID 20141303
- [Background] Atanes AC, Andreoni S, Hirayama MS, Montero-Marin J, Barros VV, Ronzani TM, Kozasa EH, Soler J, Cebolla A, Garcia-Campayo J, Demarzo MM. Mindfulness, perceived stress, and subjective well-being: a correlational study in primary care health professionals. BMC Complement Altern Med. 2015 Sep 2;15:303. doi: 10.1186/s12906-015-0823-0. PMID 26329810
- [Background] Beach MC, Roter D, Korthuis PT, Epstein RM, Sharp V, Ratanawongsa N, Cohn J, Eggly S, Sankar A, Moore RD, Saha S. A multicenter study of physician mindfulness and health care quality. Ann Fam Med. 2013 Sep-Oct;11(5):421-8. doi: 10.1370/afm.1507. PMID 24019273
- [Background] Smith SA. Mindfulness-based stress reduction: an intervention to enhance the effectiveness of nurses' coping with work-related stress. Int J Nurs Knowl. 2014 Jun;25(2):119-30. doi: 10.1111/2047-3095.12025. Epub 2014 Feb 26. PMID 24612607
- [Background] Regehr C, Glancy D, Pitts A, LeBlanc VR. Interventions to reduce the consequences of stress in physicians: a review and meta-analysis. J Nerv Ment Dis. 2014 May;202(5):353-9. doi: 10.1097/NMD.0000000000000130. PMID 24727721
- [Background] Goodman MJ, Schorling JB. A mindfulness course decreases burnout and improves well-being among healthcare providers. Int J Psychiatry Med. 2012;43(2):119-28. doi: 10.2190/PM.43.2.b. PMID 22849035
- [Background] Kemper KJ, Khirallah M. Acute Effects of Online Mind-Body Skills Training on Resilience, Mindfulness, and Empathy. J Evid Based Complementary Altern Med. 2015 Oct;20(4):247-53. doi: 10.1177/2156587215575816. Epub 2015 Mar 17. PMID 25783980